CLINICAL TRIAL: NCT04566120
Title: Detection of Streptococcus Mutans Cariogenicity by Real-time PCR in High Caries Risk Patients Using Cinnamon Extract or Chlorohexidine Mouthwashes: A Randomized Clinical Trial
Brief Title: Streptococcus Mutans Cariogenicity by Real-time PCR in High Caries Risk Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mostafa Mahmoud Mohamed Kamel El-Ghazali, Principle Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: oper131
Record Dates: First submitted 2020-09-22; First posted 2020-09-28 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Streptococcus Mutans; High Caries Risk Patients

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cinnamon extract mouthwash (Experimental): Participants will be exposed to cinnamon extract mouthwash and will be instructed to use 10 ml of cinnamon extract mouthwash 2 times per day for 1 minute; such a regimen will be continued for one month.
  Interventions: Drug: cinnamon extract mouthwash
- Chlorohexidine based mouthwash (Active Comparator): Participants will be exposed to chlorohexidine based mouthwash. and will be instructed to use 10 ml of 0.12% chlorhexidine based mouthwash 2 times per day for 1 minute; such a regimen will be continued for one month.
  Interventions: Drug: chlorohexidine based mouthwash

INTERVENTIONS:
Drug: cinnamon extract mouthwash — cinnamon extract mouthwash
  Other Names: Natural Product Mouthwash
  Arms: Cinnamon extract mouthwash
Drug: chlorohexidine based mouthwash — chlorohexidine based mouthwash
  Other Names: Synthetic Mouthwash
  Arms: Chlorohexidine based mouthwash

SUMMARY:
In patients with high caries risk, will the use of cinnamon extract or chlorohexidine based mouthwashes have an effect on the percentage of recovery and cariogenicity of Streptococcus mutans (SM) detected by real-time Polymerase Chain Reaction (PCR) over one month follow up

DETAILED DESCRIPTION:
This clinical study will be held in the clinic of conservative dentistry department, Faculty of Dentistry, Cairo University. The operator in charge will be Mostafa Mahmoud El-Ghazali. Patients will be examined and selected according to inclusion and exclusion criteria, the purpose and method of the study will be explaned to the selected patients, written informed consent will be obtained from the patients for participation in the study. In the first visit, ADA caries risk assessment model will be done. Participants will be divided into two groups according to the tested mouthwashes.

All patients will be instructed not to have breakfast and to refrain any oral hygiene measures on the day of sample collection to avoid the inﬂuence of food consumption and contamination on the composition of saliva. The patient will sit in an erect position on the dental chair and will be given paraffin block to chew. The stimulated saliva will be collected after 2 minutes of paraffin chewing in sterile containers held near the mouth. The containers will be properly labeled. The study will be carried over a period of one month, the saliva samples for each patient will be collected on the ﬁrst dental visit. These samples will be then sent to the laboratory for microbiological assessment. Patients will be provided with mouthwashes according to the tested groups and they will be instructed to use it 2 times per day for 1 minute each time and no eating or drinking permitted for a minimum of 30 minutes post rinsing. Each patient will be given the same instructions with respect to oral hygiene measures. They will be advised to continue on same diet and will be instructed not to change their dietary habits. Patients will come after 2 weeks for salivary samples collection and samples will be sent to the laboratory for microbiological assessment. After treatment continuity for another 2 weeks, patients will come for the last visit to collect the salivary samples which will be sent to the laboratory for microbiological assessment.

ELIGIBILITY:
Inclusion Criteria:

* Adults will be recruited in this study, all the volunteers participated in this experiment will be healthy looking with free medical history.
* Age range 20-50 years
* High caries risk patients according to ADA caries risk assessment model.
* High plaque index (>score 2)
* Non-smoking patients.
* Patients with normal salivary rate (0.3-0.4 ml/min).

Exclusion Criteria:

* Patients with a compromised medical history.
* Participants with low caries risk.
* Patients with severe or active periodontal disease.
* Participants with a history of allergy to any of the drugs or chemicals used in the study.
* Patients on any antibiotics during the past month
* Smoking patients.
* Patients with abnormal salivary rate.
* Pregnant female patients

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Total bacterial count | 1 month
  quantitative plating (standard plate count or SPC)n will be used to determine the number of bacteria in a culture sample. SPC reveals information on viable organisms only; bacteria colonies that are seen in the plates after incubation represent only living organisms, not dead ones.

SECONDARY OUTCOMES:
Bacterial Identification | 1 month
  Total extraction of DNA: Total plasmid DNA will be prepared. The solution will be centrifuged and then left at room temperature for few minutes for the phase separations. The aqueous phase containing DNA will be transferred to clean eppendorf.
  PCR Polymerase chain reaction: The PCR will be performed in 25µl reaction volume containing: DNA template, enzymes, primer and nuclease-free water. The tubes containing the PCR mixture will be transferred to the thermal cycler apparatus. The PCR products will be analyzed in agarose gel by electrophoresis, photographed and analyzed.
Glycosyltransferase B & D gene expression. | 1 month
  The real time PCR for relative quantification of target bacterial genes will be performed in a total volume of 20 μL using 10 µL SYBR® Premix Ex TaqTM master mix, 0.4 µL of each forward and reverse primer, 0.08 µL diluted ROX, and 2 µL of DNA template

CONTACTS AND LOCATIONS:
Overall Officials: Mostafa El-Ghazali, Principal Investigator — Assistant Lecturer
Locations (1):
- Cairo Uniuversity, Giza, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Undecided
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Expecting to have all the data by October 2022
Access Criteria: IPD through contacting the main author mostafa.elghazali@dentistrt.cu.edu.eg